CLINICAL TRIAL: NCT03255304
Title: Influence of Priming on Goal-directed and Cue-dependent Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Sabine Frank, Research Associate, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PIT_prime
Record Dates: First submitted 2017-08-14; First posted 2017-08-21 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Eating Behavior; Habits
MeSH Terms: conditions — Feeding Behavior; Habits

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- health prime (Experimental)
  Interventions: Behavioral: health mindest
- palatability prime (Experimental)
  Interventions: Behavioral: palatability mindset

INTERVENTIONS:
Behavioral: health mindest — groups be confronted with health aspects of food items
  Arms: health prime
Behavioral: palatability mindset — groups be confronted with palatability aspects of food items
  Arms: palatability prime

SUMMARY:
The current proposal aims to investigate implicit and explicit priming paradigms for changing cue-dependent and goal-directed nutritional behavior.

DETAILED DESCRIPTION:
Food choice and intake is a daily and throughout normal subject. However, for more and more people eating habits and the question of food choice are of increasing interest and in several cases even a problem. The prevalence of obesity has tripled in the last decades and it is even spoken of an obesity epidemic. Life style interventions to lose weight often fail on the long run, also because people fall back into former unhealthy eating habits. Various factors influence our daily food choice, not all of which are apparent to ourselves. Thus, food choice might be goal-directed and therefore conscious and reflective, yet in other circumstances the choice to eat something specific might be based on cue dependent processes which are automatic and thus difficult to control. Since a change in eating-behavior and long-lasting weight loss is most problematic to achieve, the current proposal aims to investigate implicit and explicit priming paradigms for changing cue-dependent and goal-directed nutritional behavior.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* currently dieting
* intolerance to provided food
* cognitive impairment

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 222 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
behavior | pre and post priming (directly before and directly after a 5 minutes priming paradigm)
  change in food choice within a Pavlovian-to-instrumental transfer task (duration of complete protocol about 45 minutes, including priming (5 minutes) and pre and post measurements)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tübingen, Tübingen, Germany